CLINICAL TRIAL: NCT00995293
Title: An Open-label, Randomized, Parallel-group, Multicenter Study of Neoadjuvant Docetaxel(Taxotere®) Plus Cisplatin Plus 5-fluorouracil Versus Neoadjuvant Cisplatin Plus 5-fluorouracil in Patients With Locally Advanced Inoperable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Taxotere (Docetaxel) New Indication: Squamous Cell Carcinoma of the Head and Neck (SCCHN) Treatment Registration Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_02557
Record Dates: First submitted 2009-09-22; First posted 2009-10-15 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel Cisplatin 5-Fluorouracil (DCF) (Experimental): 4 cycles of the following products every 3 weeks (unless disease progression/relapse or unacceptable toxicity occured or the patient refused treatment):
  * Docetaxel 60mg/m² on day 1
  * Cisplatin 75mg/m² on day 1
  * 5-FU 750mg/m²/day on day 1 to day 5
  Interventions: Drug: DOCETAXEL; Drug: CISPLATIN; Drug: 5-FLUOROURACIL
- Cisplatin 5-Fluorouracil (CF) (Experimental): 4 cycles of the following products every 3 weeks (unless disease progression/relapse or unacceptable toxicity occured or the patient refused treatment):
  * Cisplatin 75mg/m² on day 1
  * 5-FU 750mg/m²/day on day 1 to day 5
  Interventions: Drug: CISPLATIN; Drug: 5-FLUOROURACIL

INTERVENTIONS:
Drug: DOCETAXEL — Intravenous
  Arms: Docetaxel Cisplatin 5-Fluorouracil (DCF)
Drug: CISPLATIN — Intravenous
Drug: 5-FLUOROURACIL — Intravenous

SUMMARY:
The Primary Objective is to evaluate the progression-free survival after treatment with docetaxel plus cisplatin plus 5-Fluorouracil (5-FU) (DCF) in comparison with cisplatin plus 5-FU (CF) in patient with locally advanced inoperable SCCHN The Secondary Objective is to evaluate and compare the clinical response rate both before and after radiotherapy, the local symptoms, the duration of response, the time to treatment failure, the survival, the toxicity and the quality of life in the 2 study groups.

ELIGIBILITY:
Inclusion criteria:

* Tumor type: Histologically or cytologically proven squamous cell carcinoma of the head and neck (SCCHN) presenting with locally advanced disease at diagnosis. Primary tumor sites eligible are: oral cavity, oropharynx, hypopharynx and larynx.
* Extent of the disease:

  * Patients are required to have at least one measurable lesion.
  * Stage III or IV without evidence of distant metastases, according to the TNM staging system. Absence of metastases must be checked by chest X-ray (with or without Computed tomography (CT) ), abdominal ultrasound or CT in case of liver function test abnormalities, and bone scan in case of local symptoms.
  * Tumor considered as inoperable after evaluation by a multidisciplinary team. Reason for inoperability will be reported in the CRF
* World Health Organization (WHO) performance status 0 or 1
* Laboratory data:

  * Haematology:
* Neutrophil count > or = 2.0*10^9/L
* Platelet count > or = 100*10^9/L
* Hemoglobin > or = 10 g/dl (6.2 mmol/L)

  * Hepatic function:
* Total serum bilirubin < or = 1 time the upper normal limit (UNL) of the participating center
* Aspartate transaminase (ASAT/SGOT) and Alanine transaminase (ALAT/SGPT) < or = 2.5UNL
* Alkaline phosphatase < or = 5 UNL
* Patients with ASAT or ALAT > 1.5UNL associated with alkaline phosphatase >2.5UNL are not eligible for the study

  * Renal function:
* serum creatinine < or = 120µmol/L (1.4 mg/dl) if values are >120µmol/L, creatinine clearance should be > or = 60 ml/min
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, those conditions should be discussed with the patient before registration in the trial
* Patients informed consent form obtained

Exclusion criteria:

* Tumors of the nasopharynx, the nasal and paranasal cavities.
* Previous chemotherapy or radiotherapy for any reason and previous surgery for SCCHN at time of study entry.
* Prior treatment within a therapeutic clinical tria within 30 days prior to study entry
* Concurrent treatment with any other anticancer therapy
* Chronic treatment (> or = 3 months) with corticosteroids at a daily dose > or = 20mg methylprednisolone or equivalent.
* Concomitant use of drugs which could interact with 5-fluorouracil (e.g. cimetidine, allopurinol, folic or folinic acid, methotrexate and metronidazole)
* Previous or current malignancies at other sites with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years
* Symptomatic peripheral neuropathy > or = grade 2 by NCIC-CTG criteria
* Clinical altered hearing
* Pregnant, lactating women or of childbearing potential unless adequate
* with other serious illness or medical condition including but not limited to:

  * unstable cardiac disease despite treatment
  * myocardial infarction within 6 months prior to study entry
  * history of significant neurologic or psychiatric disorders including dementia or seizures
  * active uncontrolled infection
  * active peptic ulcer
  * chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to any progression event or patient death (follow-up every 3 months 1st year, then every 6 months)

SECONDARY OUTCOMES:
Overall survival | From randomization to patient death (follow-up every 3 months 1st year, then every 6 months)
Overall response rates | From randomization to any progression event or patient death (follow-up every 3 months 1st year, then every 6 months) and at the end of chemotherapy + end of radiotherapy
Duration of response | From randomization to any progression event or patient death (follow-up every 3 months 1st year, then every 6 months)
Time to treatment failure | From randomization to any progression event or patient death (follow-up every 3 months 1st year, then every 6 months) and at the end of chemotherapy + end of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mo Chen, Study Director — Sanofi
Locations (1):
- Sanofi Administrative Office, Shanghai, China